CLINICAL TRIAL: NCT05867004
Title: Blocking TNF to Potentiate the ICI-dependent Immune Awakening in Melanoma
Acronym: ATPIC
Status: Recruiting | Type: Observational
Sponsor: Institut Claudius Regaud (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: 23RT01
Record Dates: First submitted 2023-04-28; First posted 2023-05-19 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Melanoma; Immune Defect; Tumor Skin
Keywords: Melanoma; Immune checkpoint inhibitors; TNF; Resistance
MeSH Terms: conditions — Melanoma; Skin Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Blood and tumor biopsies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Cutaneous melanoma is a bad prognosis skin cancer, which can be treated with immune checkpoint inhibitors (ICI), such as anti-PD-1 (nivolumab, nivo) and anti-CTLA-4 (ipilimumab, ipi). However, about 50% of patients do not respond or relapse within 3 years post therapy induction, and immune-related adverse events (irAEs), such as colitis, are triggered and can be treated with TNF inhibitor (TNFi; ie, infliximab, inflix). The pharmacodynamic impact of TNFi on the immune and clinical responses remain to be clarified. The investigators previously demonstrated that TNFi enhance the efficacy of ICI in mouse melanoma models. Based on preclinical findings, the investigators implemented two clinical trials in advanced melanoma patients, TICIMEL and MELANFalpha. In TICIMEL, patients are concomitantly treated with TNFi [certolizumab (certo) or inflix] and ICI (ipi+nivo). In MELANFalpha, patients are treated with ICI alone. Preliminary results show both tritherapies promote systemic MART-1 specific CD8 T cell responses and that certo but not inflix may improve ICI efficacy and Th1 responses. In mouse melanoma models, TNFi enhance the response to ICI. Investigators' primary objective is to decipher how certolizumab and infliximab influence ICI-dependent anti-tumor immune responses in advanced melanoma patients. The secondary objectives are to analyse the cellular and molecular impact anti-TNF have on ICI-dependent anti-melanoma immune responses and clinical activities (irAEs and efficacy). By combining mouse and human data as well ex vivo functional assays, the investigators will dissect the impact treatments have on anti-melanoma immune responses by flow cytometry and transcriptomic analyses. The investigators expect to clarify (i) the mechanisms by which TNFi enhance ICI efficacy, (ii) identify the best TNFi to be combined with ICI in advanced melanoma patients and (iii) discover TNF-dependent biomarkers of resistance.

DETAILED DESCRIPTION:
Background and originality of the project with regards to the state of the art

Despite the tremendous breakthrough immune checkpoint inhibitors (ICI) such as anti-PD-1 and anti-CTLA-4 brought for the treatment of advanced melanoma patients, 60% of them do not respond or relapse within 5 years following treatment initiation. Severe immune-related adverse events (irAEs) are triggered upon ICI therapy, such as colitis, which can be treated with inhibitors (TNFi) of the Tumor Necrosis Factor alpha (TNF) such as infliximab. The pharmacodynamic impact of TNFi on the immune and clinical responses remains to be clarified.

Although TNF has been identified as a soluble factor able to trigger tumor necrosis in mice, the chronic production of TNF in the tumor microenvironment was shown to contribute to cancer progression. The investigators and others have shown this cancer promoting property relies on multiple mechanisms, including immune escape. For instance, the investigators showed that TNF triggers activation-induced cell death (AICD) in CD8 T cells, thereby limiting the infiltration of CD8 T cells in mouse melanoma tumors. In mouse models of melanoma, breast and colon cancers, TNFi enhance ICI (anti-PD-1, anti-CTLA-4) efficacy and reduce the severity of irAEs such as colitis. Hence, combining TNF-blocking antibodies to ICI promotes therapy efficacy and tolerance in vivo.

Investigators' unpublished data show all treatments promoted the differentiation of circulating T cells towards an effector memory phenotype (data not shown) between baseline (before treatment induction, week 0 [W0]) and week 6 (W6) post-treatment induction. They also significantly 1- Background and originality of the project with regards to the state of the art Despite the tremendous breakthrough immune checkpoint inhibitors (ICI) such as anti-PD-1 and anti-CTLA-4 brought for the treatment of advanced melanoma patients, 60% of them do not respond or relapse within 5 years following treatment initiation. Severe immune-related adverse events (irAEs) are triggered upon ICI therapy, such as colitis, which can be treated with inhibitors (TNFi) of the Tumor Necrosis Factor alpha (TNF) such as infliximab. The pharmacodynamic impact of TNFi on the immune and clinical responses remains to be clarified. Although TNF has been identified as a soluble factor able to trigger tumor necrosis in mice, the chronic production of TNF in the tumor microenvironment was shown to contribute to cancer progression. The investigatorsand others have shown this cancer promoting property relies on multiple mechanisms, including immune escape. For instance, the investigators showed that TNF triggers activation-induced cell death (AICD) in CD8 T cells, thereby limiting the infiltration of CD8 T cells in mouse melanoma tumors. In mouse models of melanoma, breast and colon cancers, TNFi enhance ICI (anti-PD-1, anti-CTLA-4) efficacy and reduce the severity of irAEs such as colitis. Hence, combining TNF-blocking antibodies to ICI promotes therapy efficacy and tolerance in vivo. Based on preclinical studies, the investigators implemented two clinical trials (TICIMEL and MELANFalpha) in advanced melanoma patients (stage IIIc/IV) treated with ICI [anti-PD-1, nivolumab (nivo) + anti-CTLA-4, ipilimumab (ipi)] in combination (TICIMEL) or not (MELANFalpha) with TNFi [certolizumab (certo) or infliximab (inflix)]. Whereas inflix is a bivalent anti-TNF chimeric IgG1 monoclonal antibody, certo is a monovalent PEGylated Fab' fragment of a humanized anti-TNF monoclonal. All patients (i.e., 92) have been enrolled between 2018 and 2021. TICIMEL (n=32) is a phase 1b clinical trial aiming at evaluating the safety and tolerability of co-administering ipi, nivo and TNFi (certo or inflix). Investigators' first data, obtained from 14 patients, indicate that both tritherapies are safe in humans, with a promising high response rate in the certo cohort. MELANFalpha (n=60) is a pilot study aiming at discovering predictive biomarkers of response/resistance to ICI. It notably shows high TNF levels are detected upon ipi/nivo treatment in plasmas from non-responders. Investigators' unpublished data show all treatments promoted the differentiation of circulating T cells towards an effector memory phenotype between baseline (before treatment induction, week 0 [W0]) and week 6 (W6) post-treatment induction. They also significantly increased the proportion of Th1 T cells in patients' blood. However, those effects were significantly amplified in the certolizumab cohort as compared to the ipi/nivo one. Accordingly, the investigators observed increased IFN-gamma plasma concentrations in the certolizumab cohort. Proportions of Th2, Th17 and Th1/17 T cells were not significantly affected by the three treatment regimens. Moreover, TNFi combination with ICI was associated with increased proportions of circulating MART-1-specific CD8 T cells. These cells mainly exhibited a central/effector memory phenotype and show increased expression of CXCR3 (Fig. 1D-F). The investigators performed CiteSeq single cell RNA sequencing (scRNAseq) on peripheral blood mononuclear cells (PBMCs) obtained before (W0) and at W6 from 4 advanced melanoma patients enrolled in each of the 3 cohorts. Signs of activation and maturation of immune responses were obvious in all patients from TICIMEL, but one, at W6. This indicates TNFi unlikely compromise the immune boost observed in patients treated with ipi/nivo. Moreover, the investigators show in a mouse melanoma model (B16Ova) whereby treatment conditions mimic that of TICIMEL and MELANFalpha (alphaPD-1+alphaCTLA-4+/- TNFi [anti-mouse TNF, clone XT3.11]), that the tritherapy increased the frequency of total tumor regressions and overall survival, as compared to the bitherapy. Mice, cured upon tritherapy, developed anti-melanoma memory responses, as evidenced by a rechallenge experiment. Understanding how TNF blockade increases the awakening of patients' anti-melanoma immune responses upon ICI and how the properties of TNFi may differentially modulate these responses is pivotal to:

* (i) get a better understanding of the cellular and molecular pathways, which need to be engaged to overcome some of the mechanisms responsible for ICI resistance.
* (ii) identify new and potentially better strategies to promote these responses.
* (iii) identify patients who might benefit the most from such therapies.

Hypothesis, main objective(s) and endpoint(s) of the project

Considering investigators' recently published and unpublished data, the investigators hypothesize that TNF blockade may promote ICI efficacy in patients. This effect may however be affected by the structural properties of the TNF blocking agent used. To evaluate this hypothesis, the investigators will compare the clinicobiological responses of patients from the TICIMEL (ipi+nivo+certo or inflix) and MELANFalpha (ipi+nivo, without TNFi) clinical trials. To clarify the molecular mechanisms by which certo and inflix differently impact on immune responses, the investigators will perform ex vivo and in vivo experiments in co-culture systems as well as in a unique mouse melanoma model, respectively.

Project plan describing the methodology and work to be performed To reach the primary and secondary objectives, the proposal is divided into three main WPs.

WP1: To decipher how certolizumab and infliximab influence the ICI-dependent systemic immune responses in advanced melanoma patients.

WP2: To analyse the impact TNFi have on ICI-dependent anti-melanoma immune responses in tumors in advanced melanoma patients. The investigators already performed immunohistochemistry (IHC) on formalin-fixed paraffin-embedded (FFPE) melanoma biopsies from patients enrolled in the first part of TICIMEL to evaluate the tumor-infiltrating leukocytes before and along therapy (CD3, CD8, CD4, FOXP3, CD68).

WP3: To analyse the impact TNFi have on ICI-dependent anti-melanoma immune responses in co-culture experiments and in mice.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion in TICIMEL clinical trial (NCT03293784),
* Inclusion in MELANFα trial (NCT03348891)

Exclusion Criteria:

* NA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with melanoma included in TICIMEL and MELANFalpha trials.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-07-03 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
To decipher how certolizumab and infliximab influence the ICI-dependent systemic immune responses in advanced melanoma patients | 36 months
  In patients from the MELANFalpha trial as well as in patients from the second phase of TICIMEL, influence of the different therapies on the capacity of circulating CD4 and CD8 T cells to produce IFNgamma, TNF and IL-17 ex vivo will be counted by flow cytometry in PBMCs.
  In patients enrolled in the second part of TICIMEL and in the ipi/nivo cohort of MELANFalpha, the evaluation of poucentage of HLA-A2 positive melanoma patients displaying circulating CD8 T cells reactive towards the tyrosinase and/or MART-1 antigens will be evaluate after staining.
  CiteSeq scRNAseq on PBMCs from patients from the 3 cohorts, including two non-responders of the ipi/nivo/certo cohort will be realise. PBMC's RNA obtained at W0 and W6 will be compared.

SECONDARY OUTCOMES:
To analyse the impact TNFi have on ICI-dependent anti-melanoma immune responses in tumors in advanced melanoma patients | 36 months
  To evaluate the tumor-infiltrating leukocytes before and along therapy (CD3, CD8, CD4, FOXP3, CD68), immunohistochemistry (IHC) on tumor samples on biopsies from patients enrolled in the second part of TICIMEL and on FFPE biopsies from MELANFalpha patients will be realised.
  To further characterize immune responses in tumors from patients enrolled in TICIMEL and MELANFalpha, RNAseq analyses on RNA extracted from pre-treatment and, when possible, matched post-treatment FFPE tumor biopsies will be performed. Differential immune signatures according to treatment and response will be assessed.
  To combine all biological and clinical data from patients by biostatistical and bioinformatic analyses. Flow cytometry, CiteSeq scRNAseq data obtained on circulating immune cells as well as IHC and RNAseq data from tumor biopsies will be combined to clinical data using machine learning methods.
To analyse the impact TNFi have on ICI-dependent anti-melanoma immune responses in co-culture experiments and in mice | 36 months
  The baseline PBMCs proliferation and the production of IFNgamma will be measured in presence of autologous CD14+ monocytes and antigenic peptides from tyrosinase or MART-1. IFNgamma plasma concentration is determined by mesoscale (pg/mL). Proliferation is measured by flow cytometry.

CONTACTS AND LOCATIONS:
Overall Officials: Bruno SEGUI, Pr, Principal Investigator — Cancer Research Center of Toulouse
Locations (1):
- Institut Claudius Regaud, Toulouse, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Larkin J, Chiarion-Sileni V, Gonzalez R, Grob JJ, Rutkowski P, Lao CD, Cowey CL, Schadendorf D, Wagstaff J, Dummer R, Ferrucci PF, Smylie M, Hogg D, Hill A, Marquez-Rodas I, Haanen J, Guidoboni M, Maio M, Schoffski P, Carlino MS, Lebbe C, McArthur G, Ascierto PA, Daniels GA, Long GV, Bastholt L, Rizzo JI, Balogh A, Moshyk A, Hodi FS, Wolchok JD. Five-Year Survival with Combined Nivolumab and Ipilimumab in Advanced Melanoma. N Engl J Med. 2019 Oct 17;381(16):1535-1546. doi: 10.1056/NEJMoa1910836. Epub 2019 Sep 28. PMID 31562797
- [Background] Brahmer JR, Lacchetti C, Thompson JA. Management of Immune-Related Adverse Events in Patients Treated With Immune Checkpoint Inhibitor Therapy: American Society of Clinical Oncology Clinical Practice Guideline Summary. J Oncol Pract. 2018 Apr;14(4):247-249. doi: 10.1200/JOP.18.00005. Epub 2018 Mar 8. No abstract available. PMID 29517954
- [Background] Chen AY, Wolchok JD, Bass AR. TNF in the era of immune checkpoint inhibitors: friend or foe? Nat Rev Rheumatol. 2021 Apr;17(4):213-223. doi: 10.1038/s41584-021-00584-4. Epub 2021 Mar 8. PMID 33686279
- [Background] Montfort A, Virazels M, Colacios C, Meyer N, Segui B. Combining TNF blockade with immune checkpoint inhibitors in patients with cancer. Nat Rev Rheumatol. 2021 Sep;17(9):577. doi: 10.1038/s41584-021-00653-8. No abstract available. PMID 34226729
- [Background] Carswell EA, Old LJ, Kassel RL, Green S, Fiore N, Williamson B. An endotoxin-induced serum factor that causes necrosis of tumors. Proc Natl Acad Sci U S A. 1975 Sep;72(9):3666-70. doi: 10.1073/pnas.72.9.3666. PMID 1103152
- [Background] Balkwill F. Tumour necrosis factor and cancer. Nat Rev Cancer. 2009 May;9(5):361-71. doi: 10.1038/nrc2628. Epub 2009 Apr 3. PMID 19343034
- [Background] Montfort A, Colacios C, Levade T, Andrieu-Abadie N, Meyer N, Segui B. Corrigendum: The TNF Paradox in Cancer Progression and Immunotherapy. Front Immunol. 2019 Oct 22;10:2515. doi: 10.3389/fimmu.2019.02515. eCollection 2019. PMID 31695705
- [Background] Bertrand F, Rochotte J, Colacios C, Montfort A, Tilkin-Mariame AF, Touriol C, Rochaix P, Lajoie-Mazenc I, Andrieu-Abadie N, Levade T, Benoist H, Segui B. Blocking Tumor Necrosis Factor alpha Enhances CD8 T-cell-Dependent Immunity in Experimental Melanoma. Cancer Res. 2015 Jul 1;75(13):2619-28. doi: 10.1158/0008-5472.CAN-14-2524. Epub 2015 May 14. PMID 25977337
- [Background] Bertrand F, Montfort A, Marcheteau E, Imbert C, Gilhodes J, Filleron T, Rochaix P, Andrieu-Abadie N, Levade T, Meyer N, Colacios C, Segui B. TNFalpha blockade overcomes resistance to anti-PD-1 in experimental melanoma. Nat Commun. 2017 Dec 22;8(1):2256. doi: 10.1038/s41467-017-02358-7. PMID 29273790
- [Background] Perez-Ruiz E, Minute L, Otano I, Alvarez M, Ochoa MC, Belsue V, de Andrea C, Rodriguez-Ruiz ME, Perez-Gracia JL, Marquez-Rodas I, Llacer C, Alvarez M, de Luque V, Molina C, Teijeira A, Berraondo P, Melero I. Prophylactic TNF blockade uncouples efficacy and toxicity in dual CTLA-4 and PD-1 immunotherapy. Nature. 2019 May;569(7756):428-432. doi: 10.1038/s41586-019-1162-y. Epub 2019 May 1. PMID 31043740
- [Background] Montfort A, Dufau C, Colacios C, Andrieu-Abadie N, Levade T, Filleron T, Delord JP, Ayyoub M, Meyer N, Segui B. Anti-TNF, a magic bullet in cancer immunotherapy? J Immunother Cancer. 2019 Nov 14;7(1):303. doi: 10.1186/s40425-019-0802-y. PMID 31727152
- [Background] Montfort A, Filleron T, Virazels M, Dufau C, Milhes J, Pages C, Olivier P, Ayyoub M, Mounier M, Lusque A, Brayer S, Delord JP, Andrieu-Abadie N, Levade T, Colacios C, Segui B, Meyer N. Combining Nivolumab and Ipilimumab with Infliximab or Certolizumab in Patients with Advanced Melanoma: First Results of a Phase Ib Clinical Trial. Clin Cancer Res. 2021 Feb 15;27(4):1037-1047. doi: 10.1158/1078-0432.CCR-20-3449. Epub 2020 Dec 3. PMID 33272982
- [Background] Balanca CC, Salvioni A, Scarlata CM, Michelas M, Martinez-Gomez C, Gomez-Roca C, Sarradin V, Tosolini M, Valle C, Pont F, Ferron G, Gladieff L, Vergez S, Dupret-Bories A, Mery E, Rochaix P, Fournie JJ, Delord JP, Devaud C, Martinez A, Ayyoub M. PD-1 blockade restores helper activity of tumor-infiltrating, exhausted PD-1hiCD39+ CD4 T cells. JCI Insight. 2021 Jan 25;6(2):e142513. doi: 10.1172/jci.insight.142513. PMID 33332284
- [Background] Atretkhany KN, Mufazalov IA, Dunst J, Kuchmiy A, Gogoleva VS, Andruszewski D, Drutskaya MS, Faustman DL, Schwabenland M, Prinz M, Kruglov AA, Waisman A, Nedospasov SA. Intrinsic TNFR2 signaling in T regulatory cells provides protection in CNS autoimmunity. Proc Natl Acad Sci U S A. 2018 Dec 18;115(51):13051-13056. doi: 10.1073/pnas.1807499115. Epub 2018 Nov 29. PMID 30498033
- [Background] Imbert C, Montfort A, Fraisse M, Marcheteau E, Gilhodes J, Martin E, Bertrand F, Marcellin M, Burlet-Schiltz O, Peredo AG, Garcia V, Carpentier S, Tartare-Deckert S, Brousset P, Rochaix P, Puisset F, Filleron T, Meyer N, Lamant L, Levade T, Segui B, Andrieu-Abadie N, Colacios C. Resistance of melanoma to immune checkpoint inhibitors is overcome by targeting the sphingosine kinase-1. Nat Commun. 2020 Jan 23;11(1):437. doi: 10.1038/s41467-019-14218-7. PMID 31974367
- [Background] Garandeau D, Noujarede J, Leclerc J, Imbert C, Garcia V, Bats ML, Rambow F, Gilhodes J, Filleron T, Meyer N, Brayer S, Arcucci S, Tartare-Deckert S, Segui B, Marine JC, Levade T, Bertolotto C, Andrieu-Abadie N. Targeting the Sphingosine 1-Phosphate Axis Exerts Potent Antitumor Activity in BRAFi-Resistant Melanomas. Mol Cancer Ther. 2019 Feb;18(2):289-300. doi: 10.1158/1535-7163.MCT-17-1141. Epub 2018 Nov 27. PMID 30482853
- [Background] Montfort A, Bertrand F, Rochotte J, Gilhodes J, Filleron T, Milhes J, Dufau C, Imbert C, Riond J, Tosolini M, Clarke CJ, Dufour F, Constantinescu AA, Junior NF, Garcia V, Record M, Cordelier P, Brousset P, Rochaix P, Silvente-Poirot S, Therville N, Andrieu-Abadie N, Levade T, Hannun YA, Benoist H, Meyer N, Micheau O, Colacios C, Segui B. Neutral Sphingomyelinase 2 Heightens Anti-Melanoma Immune Responses and Anti-PD-1 Therapy Efficacy. Cancer Immunol Res. 2021 May;9(5):568-582. doi: 10.1158/2326-6066.CIR-20-0342. Epub 2021 Mar 16. PMID 33727246
- [Background] Bilal F, Montfort A, Gilhodes J, Garcia V, Riond J, Carpentier S, Filleron T, Colacios C, Levade T, Daher A, Meyer N, Andrieu-Abadie N, Segui B. Sphingomyelin Synthase 1 (SMS1) Downregulation Is Associated With Sphingolipid Reprogramming and a Worse Prognosis in Melanoma. Front Pharmacol. 2019 Apr 30;10:443. doi: 10.3389/fphar.2019.00443. eCollection 2019. PMID 31114500